CLINICAL TRIAL: NCT06357351
Title: Comparative Evaluation of Vestibular Incision Subperiosteal Tunnel Access With Advanced Platelet-rich Fibrin and Collagen Membrane in the Treatment of Gingival Recession Defects
Brief Title: Comparison of Using Collagen Membrane and A-PRF Using VISTA Technique in Gingival Recession Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Marwa Abdelfattah Elkhamisy, Master candidate, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VISTA in gingival recession
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VISTA technique and collagen membrane (Experimental): Participants undergo periodontal surgery using the vestibular incision sub-periosteal tunnel access technique (VISTA) and collagen membrane.
  Interventions: Procedure: vestibular incision sub periosteal tunnel access ( VISTA) technique.
- VISTA technique and advanced platelet rich fibrin (Experimental): Participants undergo periodontal surgery using the vestibular incision sub-periosteal tunnel access technique (VISTA) and advanced platelet-rich fibrin (A-PRF).
  Interventions: Procedure: vestibular incision sub periosteal tunnel access ( VISTA) technique.

INTERVENTIONS:
Procedure: vestibular incision sub periosteal tunnel access ( VISTA) technique. — In comparison between the two groups, the first group uses collagen membrane and the other group uses advanced PRF using the same surgical technique (VISTA)

SUMMARY:
To assess the efficacy of minimally invasive Vestibular Incision Subperiosteal Tunnel Access (VISTA) with collagen membrane and Advanced Platelet-rich Fibrin (A-PRF) in the treatment of multiple buccal gingival recession type 1(RT1) Cairo Classification.

ELIGIBILITY:
Inclusion Criteria:

* (18-50) years old with at least 2 sites with gingival recession type (RT1) Cairo Classification (GR with no interdental attachment loss). The interdental CEJ is not detectable clinically on the labial surfaces of the teeth.
* Recession in the maxillary anterior region ≥1 mm of attached gingiva, pocket depth (PD) of <3 mm, recession depth (RD) ≥2 mm, and gingival index (GI) score ≤1.
* Systemically healthy, willing individuals with good oral hygiene and without contraindications for surgical interventions

Exclusion Criteria:

* the presence of severe systematic diseases or immunodeficiency and contraindicated with surgical interventions.
* Allergies to medicaments used in the treatment process.
* Patients with removable or fixed dentures.
* Patients with cervical abrasion, direct and indirect restorations involving the cervical areas of the maxillary anterior.
* Participants with smoking, tobacco chewing, and alcohol consumption.
* The presence of high frenal attachment and participants who had previously undergone any periodontal surgical procedure or regenerative therapy in the past 1 year at the same site of the planned treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Measuring the recession width in millimeter | baseline, 3 months and 6 months
  self-report assessment by using the UNC-15 Periodontal Probe, measured at the level of Cemento-Enamel Junction CEJ.
Measuring the recession depth in millimeter | baseline, 3 months and 6 months
  self-report assessment by using the UNC-15 Periodontal Probe, measured from the cemento-enamel junction CEJ to the free gingival junction.
Measuring the width of keratinized gingiva in millimeter | baseline, 3 months and 6 months
  self-report assessment by using the UNC-15 Periodontal Probe. measured from the free gingiva margin to the mucogingival junction.
Mean of root coverage | baseline, and 6 months
  was measured by the following formula:. Mean root coverage formula: (pre-operative recession depth - post-operative recession depth)/(pre-operative recession depth ) ×100

SECONDARY OUTCOMES:
Measuring the probing depth | baseline, 3 months and 6 months
  self-report assessment by using the UNC-15 Periodontal Probe. Measured from the free gingival margin to the base of the sulcus.
Measuring the plaque index | baseline, 3 months and 6 months
  According to Silness and Leo, this index determines the thickness of the plaque along the gingival margin. possible score range from 0 (no plaque) to 1 ( thin plaque located at gingival margin only detected by periodontal probe), 2 ( moderate plaque thickness detected by naked eye located at gingival margin), and 3 ( abundant plaque thickness at gingival margin and interproximal area)
Measuring the gingival index | baseline, 3 months and 6 months
  According to Silness and Leo, this index determines the description of the gingiva of examined teeth. possible score range from 0 (normal gingiva) to 1 (mild inflammation; slight erythema; no bleeding.) / 2 (moderate inflammation; erythema and bleeding on probing) or 3 (severe inflammation; severe erythema, swelling, and spontaneous bleeding).
Clinical attachment level | baseline, 3 months and 6 months
  self-report assessment by using the UNC-15 Periodontal Probe, measured from the cemento-enamel junction to the base of the pocket.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Egypt

REFERENCES:
- [Derived] Abdelhaleem M, Saleh W, Elmeadawy S. Treatment of gingival recession with vestibular incision subperiosteal tunnel access and advanced platelet-rich fibrin. BMC Oral Health. 2025 Jan 14;25(1):63. doi: 10.1186/s12903-024-05398-w. PMID 39806320